CLINICAL TRIAL: NCT00525538
Title: Evaluation Conformal Radiotherapy for Gynecologic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Model: Parallel | Masking: None
Other Study IDs: IUCMFRO-07
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2007-09-05 (Estimated); Status verified 2007-08

CONDITIONS: Radiation Therapy
MeSH Terms: interventions — Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: conformal radiotherapy

SUMMARY:
The purpose of this study is comparision conformal radiotherapy for gynecologic cancer

ELIGIBILITY:
Inclusion Criteria:

* Gynecologic cancer

Exclusion Criteria:

* Metastases

Sex: Female
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: filiz munzuroglu, Principal Investigator — Cerrahpasa Medical Faculty Department of Radiation Oncology
Locations (1):
- Cerrahpasa Medical Faculty Department of Radiation Oncology, Istanbul, Fatih, Turkey (Türkiye)